CLINICAL TRIAL: NCT01643785
Title: Additive Effect of Endonase on the Efficacy of Bismuth-containing Quadruple Therapy as Second-line Treatment for Helicobacter Pylori Infection
Brief Title: Additive Effect of Endonase on Eradication Rate of Second Line Therapy for HP Infection
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Chuncheon Sacred Heart Hospital (Other)
Responsible Party: Principal Investigator, Yeonsoo Kim, Assistant Professor, Chuncheon Sacred Heart Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSHH Endonase2
Record Dates: First submitted 2012-07-11; First posted 2012-07-18 (Estimated); Last update posted 2014-01-22 (Estimated); Status verified 2014-01

CONDITIONS: Helicobacter Pylori Infection
Keywords: therapeutic efficacy endonase addictive effect

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- with Endonase (Experimental): Second-line quadruple therapy [PPI(pantoprazole 40mg, lansoprazole 30mg, esomeprazole 40mg, rabeprazole 20mg, omeprazole 20mg) Bid, tetracycline 500 mg QID, metronidazole 500mg Tid, tripotassium dicitrate bismuthate 300mg QID] plus 20,000 units of pronase (endonase), BID for 7 days
  Interventions: Drug: Second-line quadruple therapy with endonase
- without Endonase (No Intervention): Second-line quadruple therapy [PPI(pantoprazole 40mg, lansoprazole 30mg, esomeprazole 40mg, rabeprazole 20mg, omeprazole 20mg) Bid, tetracycline 500 mg QID, metronidazole 500mg Tid, tripotassium dicitrate bismuthate 300mg QID] for 7 days

INTERVENTIONS:
Drug: Second-line quadruple therapy with endonase — Compare Second-line quadruple therapy w/o pronase (endonase)
  Other Names: Brand name: Endonase
  Arms: with Endonase

SUMMARY:
Endonase, a kind of protease, is known to cause both extensive degradation of mucins and a reduction in mucus viscosity. As part of the search for more effective forms of therapy against H. pylori when it colonizes not only the surface of the surface mucosal cells but also the surface mucous gel layer covering the mucosal surface of the stomach. The investigators decided to investigate whether or not endonase might have additive effect of pronase on the efficacy of the second-line eradication therapy against Helicobacter pylori.

ELIGIBILITY:
Inclusion Criteria:

Patients with 18 years or more of age AND Patients who failed the standard proton pump inhibitor-based triple therapy for H. pylori

Exclusion Criteria:

1. Patients Under 18 years, OR
2. Patients with active peptic ulcer, OR
3. Pregnant or Breast feeding women, OR
4. Patients with gastric malignancy, OR
5. Patients with a history of drug allergy or hypersensitivity, OR
6. Patients with severe renal, liver, or heart diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-06; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Eradication rate | 4 weeks
  Intention-to-treat analysis and per-protocol analysis to compare the eradication rate of the bismuth-containing quadruple therapy plus endonase as the second-line treatment with that of the bismuth-containing quadruple therapy

SECONDARY OUTCOMES:
Number of participants with adverse events | 4 weeks
  Difference in the number of participants with adverse events between patients receiving bismuth-containing quadruple therapy plus endoase as the second-line treatment for H. pylori and patients receiving only bismuth-containing quadruple therapy
Number of participants taking over 85% of medicine | 4 weeks
  Difference in the number of participants taking over 85% of medicine between patients receiving bismuth-containing quadruple therapy plus endoase as the second-line treatment for H. pylori and patients receiving only bismuth-containing quadruple therapy

CONTACTS AND LOCATIONS:
Overall Officials: JinBong Kim, MD, Principal Investigator — Chuncheon Sacred Heart Hospital
Locations (1):
- Chuncheon Sacred Heart Hospital, Chuncheon, Gangwon-do, South Korea